CLINICAL TRIAL: NCT01189487
Title: A Multicenter, Unblinded, Non-Comparative Study Of Unasyn-S 12 G/Day Evaluating The Safety And Efficacy In Japanese Adult Subjects With Community Acquired Pneumonia
Brief Title: The Study of Unasyn-S 12g/Day for Community Acquired Pneumonia (CAP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A9231001
Record Dates: First submitted 2010-08-16; First posted 2010-08-26 (Estimated); Results first posted 2012-05-18 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Pneumonia, Bacterial
Keywords: ampicillin sodium/sulbactam sodium; Unasyn-S; community acquired pneumonia; bacterial pneumonia
MeSH Terms: conditions — Pneumonia, Bacterial; Community-Acquired Pneumonia | interventions — Ampicillin; Sulbactam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ampicillin sodium/sulbactam sodium (Experimental): ampicillin sodium/sulbactam sodium 12g/day (3 g four times a day) IV
  Interventions: Drug: ampicillin sodium/sulbactam sodium

INTERVENTIONS:
Drug: ampicillin sodium/sulbactam sodium — ampicillin sodium/sulbactam sodium is administered 12g/day (3 g four times a day) intravenously for 3 to 14 days
  Other Names: Unasyn-S

SUMMARY:
Unasyn-S 12g/day (3 g four times a day) is the commonly used dosage depending on the severity for US, EU, China, Taiwan and Korea for over 20 years, however, Unasyn-S 12g/day has not yet been approved in Japan. The purpose of this trial is to evaluate the clinical efficacy and safety in Japanese adult subjects with community acquired pneumonia receiving ampicillin sodium/sulbactam sodium, 12g/day (3 g four times a day ) IV.

ELIGIBILITY:
Inclusion Criteria:

* 16 years of age or older.
* Patients who were diagnosed as moderate to severe community acquired pneumonia requiring initial intravenous therapy and hospitalization.

Exclusion Criteria:

* Known or suspected hypersensitivity or intolerance to ampicillin sodium/sulbactam sodium, other penicillins, or cephems.
* Hepatic dysfunction [Aspartate Aminotransferase(AST), Alanine Aminotransferase (ALT), total bilirubin > 3 times upper limit of normal range values].
* Severe renal dysfunction (creatinine clearance < 30 ml/min).
* Severe underlying disease; patients in which drug clinical evaluation is difficult because of confounding diseases.

Ages: 16 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- Japan (22):
  - Tosei General Hospital, Seto-shi, Aichi-ken
  - Fukuoka Sanno Hospital, Fukuoka, Fukuoka
  - National Hospital Organization Kokura Medical Center, Kitakyushu, Fukuoka
  - University of Occupational and Environmental Health, Kitakyushu, Fukuoka
  - Nagata Hospital, Yanagawa, Fukuoka
  - National Hospital Organization Asahikawa Medical Center, Asahikawa, Hokkaido
  - National Hokkaido Medical Center, Sapporo, Hokkaido
  - National Hospital Organization Himeji Medical Center, Himejishi, Hyōgo
  - KKR Takamatsu Hospital, Takamatsu, Kagawa-ken
  - Nippon Koukan Hospital, Kawasaki, Kanagawa
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama, Kanagawa
  - National Hospital Organization Kochi National Hospital, Kochi, Kochi
  - National Hospital Organization Kumamoto Saishyunsou Hospital, Koushi-shi, Kumamoto
  - Saiseikai Kumamoto Hospital, Kumamoto, Kumamoto
  - Saka General Hospital/Respiratory, Shiogama, Miyagi
  - National Hospital Organization Matsumoto Medical Center Chushin Matsumoto Hospital, Matsumoto, Nagano
  - Japanese Red Cross Nagasaki Genbaku Isahaya Hospital, Isahaya, Nagasaki
  - Nagasaki University School of Medicine, Nagasaki, Nagasaki
  - National Hospital Organization Minami-Okayama Medical Center, Tsukubo-gun, Okayama-ken
  - National Hospital Organization Ureshino Medical Center, Ureshino-shi, Saga-ken
  - Sekishinkai Sayama Hospital, Sayama, Saitama
  - National Hospital Organization Tenryu National Hospital, Hamamatsu, Shizuoka

REFERENCES:
- [Derived] Kohno S, Tateda K, Mikamo H, Kadota J, Niki Y, Itamura R. Efficacy and safety of intravenous sulbactam/ampicillin 3 g 4 times daily in Japanese adults with moderate to severe community-acquired pneumonia: a multicenter, open-label, uncontrolled study. J Infect Chemother. 2015 Mar;21(3):182-8. doi: 10.1016/j.jiac.2014.11.006. Epub 2014 Nov 20. PMID 25533886
- [Derived] Soto E, Shoji S, Muto C, Tomono Y, Marshall S. Population pharmacokinetics of ampicillin and sulbactam in patients with community-acquired pneumonia: evaluation of the impact of renal impairment. Br J Clin Pharmacol. 2014 Mar;77(3):509-21. doi: 10.1111/bcp.12232. PMID 24102758
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9231001&StudyName=The%20Study%20of%20Unasyn-S%2012g/day%20for%20Community%20Acquired%20Pneumonia%20%28CAP%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Ampicillin Sodium/Sulbactam Sodium: Intravenous ampicillin sodium/sulbactam sodium 3 g four times a day (12 g/day) for 3 to 14 days
Period: Overall Study
Arm/Group | Ampicillin Sodium/Sulbactam Sodium
Started | 47 (Treated participants)
Completed | 44
Not Completed | 3
Not completed — Lack of Efficacy | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ampicillin Sodium/Sulbactam Sodium
Number analyzed (Participants) | 47
Age Continuous [Mean (Standard Deviation); unit: years] | 62.3 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Clinical Response, Data Review Committee Assessment)
Description: Response rate was calculated from the following formula, "the number of participants assessed as effective" over "total participants excluding ones assessed as indeterminate" multiplied by 100.
Time Frame: End of treatment, Test of cure (7 days after End of treatment), Long term follow up (7 days after Test of cure)
Population: Clinical per protocol set consisted of all participants who received at least one dose, have no significant violation of protocol, and underwent prescribed evaluations during the observation period. No imputation was used for missing data. "n" in the Measure Values means total participants EXCLUDING ones assessed as indeterminate.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ampicillin Sodium/Sulbactam Sodium
Number analyzed (Participants) | 40
percentage of participants
  End of treatment (n=39) | 97.4 [86.5 to 99.9]
  Test of cure (n=37) | 94.6 [81.8 to 99.3]
  Long term follow up (n=36) | 94.4 [81.3 to 99.3]

2. Secondary Outcome: Response Rate (Clinical Response, Investigator Assessment)
Description: as for outcome 1
Time Frame: End of treatment, Test of cure (7 days after End of treatment), Long term follow up (7 days after Test of cure)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ampicillin Sodium/Sulbactam Sodium
Number analyzed (Participants) | 40
percentage of participants
  End of treatment (n=40) | 100.0 [91.2 to 100.0]
  Test of cure (n=38) | 100.0 [90.7 to 100.0]
  Long term follow up (n=34) | 100.0 [89.7 to 100.0]

3. Secondary Outcome: The Tendency Toward Clinical Improvement (Investigator Assessment)
Description: The number of participants who showed tendency toward clinical improvement based on the assessment of temperature, white blood cell count, C-reactive protein, clinical symptoms on Day 4 and was determined to continue the treatment.
Time Frame: Day 4
Population: Clinical per protocol set consisted of all participants who received at least one dose, have no significant violation of protocol, and underwent prescribed evaluations during the observation period. No imputation was used for missing data.
Measure: Number; unit: percentage of participants
Arm/Group | Ampicillin Sodium/Sulbactam Sodium
Number analyzed (Participants) | 40
percentage of participants | 100.0

4. Secondary Outcome: Eradication Rate (Bacteriological Response, Data Review Committee Assessment)
Description: Eradication Rate was calculated from the following formula, "the number of participants assessed as eradication, presumed eradication or microbial substitution" over "total participants excluding ones assessed as indeterminate" multiplied by 100. Microbial substitution means the appearance of new pathogens other than the original pathogens in a specimen from the same location with signs and symptoms of infection after the original pathogens were eradicated by treatment.
Time Frame: Day 4, End of treatment, Test of cure (7 days after End of treatment), Long term follow up (7 days after Test of cure)
Population: Bacteriologic per protocol set consisted of all participants in the clinical per protocol set in whom bacterial pathogens were identified at baseline. No imputation was used for missing data. "n" in the Measure Values was the total participants EXCLUDING ones assessed as indeterminate.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ampicillin Sodium/Sulbactam Sodium
Number analyzed (Participants) | 28
percentage of participants
  Day 4 (n=24) | 100.0 [85.8 to 100.0]
  End of treatment (n=25) | 96.0 [79.6 to 99.9]
  Test of cure (n=24) | 91.7 [73.0 to 99.0]
  Long term follow up (n=21) | 95.2 [76.2 to 99.9]

5. Secondary Outcome: Eradication Rate (Bacteriological Response, Investigator Assessment)
Description: Eradication Rate was calculated from the following formula, "the number of participants assessed as eradication , presumed eradication or microbial substitution" over "total participants excluding ones assessed as indeterminate" multiplied by 100. Microbial substitution means the appearance of new pathogens other than the original pathogens in a specimen from the same location with signs and symptoms of infection after the original pathogens were eradicated by treatment.
Time Frame: Day 4, End of treatment, Test of cure (7 days after End of treatment), Long term follow up (7 days after Test of cure)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentageof participants
Arm/Group | Ampicillin Sodium/Sulbactam Sodium
Number analyzed (Participants) | 28
percentageof participants
  Day 4 (n=23) | 95.7 [78.1 to 99.9]
  End of treatment (n=24) | 100.0 [85.8 to 100.0]
  Test of cure (n=23) | 95.7 [78.1 to 99.9]
  Long term follow up (n=19) | 100.0 [82.4 to 100.0]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Ampicillin Sodium/Sulbactam Sodium
Serious Adverse Events (participants affected / at risk) | 1/47
Other Adverse Events (participants affected / at risk) | 19/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ampicillin Sodium/Sulbactam Sodium (N=47)
Pneumonia (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ampicillin Sodium/Sulbactam Sodium (N=47)
Constipation (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 3
Pyrexia (General disorders) | 2
Nasopharyngitis (Infections and infestations) | 3
Alanine aminotransferase increased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 6
Blood alkaline phosphatase increased (Investigations) | 4
Gamma-glutamyltransferase increased (Investigations) | 3
Headache (Nervous system disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.